CLINICAL TRIAL: NCT04296903
Title: Post-approval Registry Study to Evaluate the Continued Safety and Probable Benefit of the MID-C System for 5 Years Post-Implantation in Adolescent Idiopathic Scoliosis (AIS)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Apifix (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MID-C-AIS-03-18
Record Dates: First submitted 2020-03-01; First posted 2020-03-05 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Adolescent Idiopathic Scoliosis

STUDY DESIGN:
Intervention Model Description: Prospective Registry, multi center, single arm, non-randomized, new enrollment cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- MID-C treatment (Experimental)
  Interventions: Device: MID-C System

INTERVENTIONS:
Device: MID-C System — Minimal invasive deformity correction system for the treatment of AIS

SUMMARY:
The ApiFix MID-C System is a unidirectional expandable rod, designed to be connected unilaterally to the spine via 2 anchor points on the concave side of a scoliotic deformity above and below the apex of the major curvature to treat adolescent idiopathic scoliosis. The MID-C System is designed to act as an internal brace. Patients implanted with the device in the US within 2 years of FDA's approval of H17001 should be enrolled in the study. A minimum number of 200 patients will be enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent Idiopathic Scoliosis classified as Lenke Type 1 or Type 5 curves;
* Cobb angle between 35-60 degrees (inclusive);
* Flexible curve that that reduces to ≤ 30 degrees on lateral side-bending radiographs or as evident by traction x-ray;
* Kyphosis angles of ≤ 55 degrees measured from T5 to T12;
* Appropriate candidate for posterior surgical approach;
* Patient has good general health;
* Patient has no known hypersensitivity or allergies to titanium;
* Patient's guardian signs a written informed consent form (ICF).

Exclusion Criteria:

* Any type of non-idiopathic scoliosis;
* Any main thoracic deformity that includes vertebral levels and cranial including to T2;
* Known history of existing malignancy, or any systemic or local infection;
* Spinal cord abnormalities that require treatment;
* Known neurological deficit (defined as motor grade < 5/5);
* Known poor bone quality defined as T score -1.5 or less;
* For female Patient, pregnancy;
* Previous spine surgery that would prevent the successful performance of the MID-C system ;
* Active systemic disease, such as AIDS, HIV, or active infection;
* Active infection or the skin is compromised at the surgical site;
* Systemic disease that would affect the Patient's welfare or overall outcome of the study.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2020-05-31 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Maintenance of major Cobb angle ≤ 40° 5 years post-surgery | 5 years
  Spinal Cobb angle will be measured at 5 years post op. the percent of patients with Cobb angle ≤ 40° 5 years post-surgery will be calculated

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Rady Children's Hospital, San Diego, California
  - Wolfson children's hospital, Jacksonville, Florida
  - Wellstar, Atlanta, Georgia
  - Riley Children's Health, Indianapolis, Indiana
  - Children's Mercy Hospital, Kansas City, Kansas
  - Mayo Clinic, Rochester, Minnesota
  - Univ. of Mississippi Medical Center (UMMC), Jackson, Mississippi
  - Women and Children's Hospital - University of Missouri Health Care, Columbia, Missouri
  - Shriners Hospitals for Children, St Louis, Missouri
  - Mount Sinai hospital, New York, New York
  - Rainbow babies and children, Cleveland, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - Avera Health, Sioux Falls, South Dakota
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No